CLINICAL TRIAL: NCT04456192
Title: Effects of an Indoor Cycling Program on Cardio-Metabolic Factors in Women With Obesity and Normal Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Marzena Ratajczak, assistant professor, Poznan University of Physical Education
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PoznanUPhyEd no. 2
Record Dates: First submitted 2020-06-24; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Obesity; Dyslipidemias; Hypertension; Type 2 Diabetes; Endothelial Dysfunction
Keywords: obesity; indoor cycling; interval physical training; cardio-metabolic factors
MeSH Terms: conditions — Obesity; Dyslipidemias; Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study was designed as a prospective trial where two similar groups of women only differing in body mass participate in the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women with Obesity (Experimental): 23 healthy, obese (BMI ≥ 30 kg/m2; waist circumference > 80) women, aged 34-62, screened at the outpatient clinic of the Department of Internal Medicine, Metabolic Disorders, and Hypertension, University of Medical Sciences, Poznań, Poland were enrolled based on the inclusion criteria and the willingness to participate in the research.
  Interventions: Behavioral: Indoor Cycling Interval Exercise Training
- Normal-weight Women (Active Comparator): 8 healthy, normal-weight (≤ 24.9 and ≥ 18.5 kg/m2) women, aged 34-62 were enrolled to intervention from the announcement.
  Random selection for groups was not applicable due to the planned body mass difference in the studied groups.
  Interventions: Behavioral: Indoor Cycling Interval Exercise Training

INTERVENTIONS:
Behavioral: Indoor Cycling Interval Exercise Training — The 3-month intervention consisted of a physical exercise program involving three indoor cycling sessions per week, with a total of 36 training sessions. Subjects exercised on cycle ergometers Schwinn® Evolution® (Schwinn Bicycle Company, Boulder, Colorado, USA). Each session lasted approximately 55 minutes. Training sessions consisted of a 5-min low-intensity warm-up (cycling at 50-65% of maximum heart rate (HRmax)), 40 min of main training at an intensity of 65-95% of HRmax, 5 min of non-weight-bearing cycling, finishing with 5 min of low-intensity cool-down stretching and breathing exercises.
  Main part of the training was interval. Each exercise session consisted of 3 to 4 high intensity intervals with intensity exceeding 80% of HRmax, often reaching anaerobic threshold. High intensity intervals lasted approximately 4-minutes and were interspersed by recovery periods at 65-80% of HRmax.
  Other Names: Spinning Interval Physical Training

SUMMARY:
The aim of the research is to (1) evaluate the potential clinical effectiveness and biological mechanisms of indoor cycling in the treatment of obesity and (2) provide-up-to-date evidence on the impact of indoor cycling in reducing cardiovascular disease (CVD) risk factors, namely, hypertension, dyslipidemia, type 2 diabetes, endothelial dysfunction. We hypothesize that IC training, can be a good stimulus to mitigate cardiovascular risk factors in women with obesity and to improve values of the examined indicators towards that occurring in women with normal body weight.

The study was designed as a prospective exercise intervention trial. The study involved women with obesity (OW) and women with normal body weight (NW). Both study groups underwent the same 3-month physical training program. Outside the implemented program, all participants were instructed to maintain their normal physical activity, diet and not to use any dietary supplements. Dietary intake was assessed using interviews conducted at baseline and after completion of the trial. The amount of nutrients in participant's daily diet was processed and evaluated using a dietetics computer program. The intake of nutrients, total caloric intake during the study were constant in both groups. Anthropometric parameters, blood pressure and physical capacity were measured and blood samples were taken at baseline and after completion of the physical training program.

The study involved 31 obese or normal weight women aged 34-62. A total of 23 women with obesity (body mass index (BMI) ≥ 30 kg/m2; waist circumference > 80 cm) registered and screened from among 163 women at the outpatient clinic of the Department of Internal Medicine, Metabolic Disorders, and Hypertension, University of Medical Sciences, Poznań, Poland were enrolled to OW group. The NW group consisted of 8 healthy women from the announcement (BMI ≤ 24.9 and ≥ 18.5 kg/m2).

Informed consent was obtained from all participants, and the study was approved by the Ethics Committee of Poznan University of Medical Sciences (case no. 1077/12; supplement no. 753/13). The study conformed to all ethical issues included in the Helsinki Declaration.

The 3-month intervention consisted of a physical exercise program involving three indoor cycling sessions per week, with a total of 36 training sessions. Subjects exercised on cycle ergometers Schwinn® Evolution® (Schwinn Bicycle Company, Boulder, Colorado, USA). Each session lasted approximately 55 minutes. Training sessions consisted of a 5-min low-intensity warm-up (cycling at 50-65% of maximum heart rate (HRmax)), 40 min of main training at an intensity of 65-95% of HRmax, 5 min of non-weight-bearing cycling, finishing with 5 min of low-intensity cool-down stretching and breathing exercises.

Main part of the training was interval. Each exercise session consisted of 3 to 4 high intensity intervals with intensity exceeding 80% of HRmax, often reaching anaerobic threshold. High intensity intervals lasted approximately 4-minutes and were interspersed by recovery periods at 65-80% of HRmax.

HR during sessions was monitored with a Suunto Fitness Solution® device (Suunto, Vantaa, Finland). To ensure that assigned exercise intensities were obtained, the average per cent of the maximum heart rate during the entire training session was obtained from the device Blood samples for biochemical analyses were taken from a basilic vein, after overnight 12-hour fasting. In the serum samples, parameters were measured using commercially available enzyme-linked immunoassays.

Both before and after the whole training programme, the following measurements were made: body weight and height, BMI, waist and hip circumference, WHR, body composition (DXA), total-body skeletal muscle mass index, graded exercise test, isokinetic muscle strength of knee flexors and extensors, exercise and resting blood pressure, and the heart rate. Vascular endothelial function indices (eNOS, VEGF, TBARS and TAS) as well as TCH, LDL-C, HDL-C, TG, oxLDL and CRP of venous blood were determined.

A sample size was determined according to changes in VO2 peak. A total of 6 subjects in OW group and 7 subjects in NW group was calculated to yield at least 80% power of detecting an intervention effect as statistically significant at the 0.05 α level.

DETAILED DESCRIPTION:
Anthropometric measurements were conducted with the subjects wearing light clothing and no shoes. Weight was measured to the nearest 0.1 kg and height to the nearest 0.5 cm. BMI was calculated as weight divided by height squared (kg/m2 ). Obesity was defined as BMI ≥ 30 kg/m2. Waist circumference (cm) was measured at the level of the iliac crest at the end of normal expiration. Hip circumference was measured at the maximum protuberance of the buttocks. Waist and hip circumferences were measured to the nearest 0.5 cm. Waist-to-hip ratio (WHR) was calculated as waist circumference divided by hip circumference. Index of central obesity (ICO) was calculated as waist circumference (cm) divided by height (cm) (Parikh, et al., 2012).

Body composition analysis was assessed using DXA (GE Healthcare Lunar Prodigy Advance; GE Medical Systems, Milan, Italy). The subjects were instructed not to make any intense physical effort in the 24h prior to the examination. The subjects were given complete instructions on the examination procedure. They wore cotton T-shirt, shorts, and socks and lay on the DXA table supine and motionlessly during the testing procedure. They were instructed to remove all metal, rubber, and plastic objects that might affect the X-ray beam. The same well-trained laboratory technician positioned the subjects, performed the scans, and executed the analysis according to the operator's manual, using the standard analysis protocol. Total body fat mass and lean body mass were determined using standard scan mode (in case of moderately obese subjects) or thick scan mode (in case of extremely obese subjects); the absorbed dose of radiation was 0.4 μGy and 0.8 μGy, respectively.

To determine the subjects' physical capacity, a Graded Exercise Test (GXT) was performed on an electronically braked cycle ergometer (Kettler ® DX1 Pro, Kettler, Ense, Germany). GXT began at a work rate of 25 W (60 rev/min). The work rate was incremented by 25 W every 2 min until the subject could no longer maintain the required pedal cadence. Each test lasted 4-14.5 min, depending on age and aerobic fitness status. The exercise tests were conducted between 8: 00 and 12: 00 a.m. in an air-conditioned laboratory, 2 h after consuming a light breakfast. Expired gases, minute ventilations (Ve), and heart rate (HR) during GXT were monitored continuously with an automated system (Oxycon Mobile ® ; Viasys Healthcare, Hoechberg, Germany). Oxygen intake (VO 2 ) and carbon dioxide output (VCO 2 ) was measured breath-by-breath and averaged over 15-second periods. Before each trial, the system was calibrated according to the manufacturer's instructions. Peak VO2 was defined as the highest 15-second averaged VO 2 obtained during the final exercise load on the test. HR peak (bpm) was measured as the highest 15-second average value in the test. To determine ventilatory threshold (VT), the V-slope method was administered using computerized regression analysis on the slopes of the CO 2 output versus O2 uptake plot, which detects the beginning of the excess CO 2 output generated from the buffering of H +. The method involves analyzing the behavior of VCO 2 as a function of VO 2 during GXT with a consequent increase in VCO 2 . This results in a transition in the relationship between VCO 2 and VO 2 . The software supplied by Viasys Healthcare was used, supported with a visual inspection on the part of an experienced researcher. As a secondary method, the ventilatory equivalent method (VEQ method) was employed and the point at which the equivalent for oxygen (VE/VO 2 ) increased without a concomitant rise in the equivalent for carbon dioxide (VE/VCO 2 ) was detected. The VT was expressed as a heart rate (HR VT ).

Exercise blood pressure was measured during a GXT using a digital electronic tensiometer (model 705IT TM, Omron Corporation, Kyoto, Japan). The measurement was taken during maximal work rate. Exercise HR was measured as the highest 15-second average value in the GXT. Resting blood pressure was measured fasting in the morning hours, in a sitting position with the legs uncrossed and the back and arm supported. Resting HR was measured under the same conditions, using auscultation of the heart by stethoscope. Regular or large adult cuffs were used, depending on the patient's arm circumference.

ELIGIBILITY:
Inclusion Criteria:

Initial inclusion criteria for both study groups were as follows: age: 30 to 65 years and stable body weight in the month prior to the trial (permissible deviation ± 1 kg).

For Women with Obesity Group: BMI ≥ 30 kg/m2; waist circumference > 80 cm. For Normal-weight Womeng Group: BMI ≤ 24.9 and ≥ 18.5 kg/m2

Exclusion Criteria for both study groups were as follows:

* secondary form of obesity and/or secondary form of hypertension;
* diabetes mellitus;
* history of coronary artery disease;
* stroke;
* congestive heart failure;
* clinically significant arrhythmias or conduction disorders;
* malignancy;
* poorly controlled hypertension (SBP > 140 mmHg and/or DBP > 90 mmHg), and/or modifications to antihypertensive treatment;
* lipid disorders requiring the implementation of drug treatment;
* clinically significant abnormalities in liver, kidney or thyroid gland function;
* clinically significant acute or chronic inflammatory process within the respiratory, digestive or genitourinary tracts, or the oral cavity, pharynx or paranasal sinuses; or, presence of connective tissue disease or arthritis;
* history of infection within the month prior to the study;
* nicotine, alcohol or drug abuse;
* and / or any other condition which, according to the researchers, would cause that participation would be detrimental to the participant or would prevent, limit or interfere with the results of the study.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) and triglycerides (TG) [mmol/l] | At baseline
  Dimension Flex Reagent Cartridge
Total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) and triglycerides (TG) [mmol/l] | After three months of physical training
  Dimension Flex Reagent Cartridge
Human anti-oxidized low density lipoprotein antibody (OLAb) [U/L] | At baseline
  ELISA
Human anti-oxidized low density lipoprotein antibody (OLAb) [U/L] | After three months of physical training
  ELISA
Blood total antioxidant capacity (TAC) [mmolCRE/l] | At baseline
  ELISA
Blood total antioxidant capacity (TAC) [mmolCRE/l] | After three months of physical training
  ELISA
Thiobarbituric acid reactive substances (TBARS) [μmol/l] | At baseline
  ELISA
Thiobarbituric acid reactive substances (TBARS) [μmol/l] | After three months of physical training
  ELISA
Activity of endothelial nitric oxide synthase (eNOS) [ng/ml] | At baseline
  ELISA
Activity of endothelial nitric oxide synthase (eNOS) [ng/ml] | After three months of physical training
  ELISA
Vascular endothelial growth factor (VEGF) [pg/ml] | At baseline
  ELISA
Vascular endothelial growth factor (VEGF) [pg/ml] | After three months of physical training
  ELISA
C-reactive protein concentration (CRP) [mg/l] | At baseline
  ELISA
C-reactive protein concentration (CRP) [mg/l] | After three months of physical training
  ELISA

SECONDARY OUTCOMES:
Body mass [kg] | At baseline
Body mass [kg] | After three months of physical training
Body height, waist circumference, hip circumference [cm] | At baseline
Body height, waist circumference, hip circumference [cm] | After three months of physical training
Body composition | At baseline
  Dual-energy X-ray Absorptiometry
Body composition | After three months of physical training
  Dual-energy X-ray Absorptiometry
Peak oxygen uptake (VO2 peak) [ml•min-1•kg-1] | At baseline
  Graded Exercise Test (GXT) with an automated system Oxycon Mobile ®
Peak oxygen uptake (VO2 peak) [ml•min-1•kg-1] | After three months of physical training
  Graded Exercise Test (GXT) with an automated system Oxycon Mobile ®
Resting heart rate [bpm], Peak heart rate [bpm], Ventilatory threshold heart rate [bpm], | At baseline
Resting heart rate [bpm], Peak heart rate [bpm], Ventilatory threshold heart rate [bpm], | After three months of physical training
Resting SBP [mmHg], Resting DBP [mmHg], Exercise SBP [mmHg], Exercise DBP [mmHg] | At baseline
Resting SBP [mmHg], Resting DBP [mmHg], Exercise SBP [mmHg], Exercise DBP [mmHg] | After three months of physical training

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Physical Education, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bianco A, Bellafiore M, Battaglia G, Paoli A, Caramazza G, Farina F, Palma A. The effects of indoor cycling training in sedentary overweight women. J Sports Med Phys Fitness. 2010 Jun;50(2):159-65. PMID 20585293
- [Background] Chavarrias M, Carlos-Vivas J, Collado-Mateo D, Perez-Gomez J. Health Benefits of Indoor Cycling: A Systematic Review. Medicina (Kaunas). 2019 Aug 8;55(8):452. doi: 10.3390/medicina55080452. PMID 31443139
- [Background] Damaso AR, da Silveira Campos RM, Caranti DA, de Piano A, Fisberg M, Foschini D, de Lima Sanches P, Tock L, Lederman HM, Tufik S, de Mello MT. Aerobic plus resistance training was more effective in improving the visceral adiposity, metabolic profile and inflammatory markers than aerobic training in obese adolescents. J Sports Sci. 2014;32(15):1435-45. doi: 10.1080/02640414.2014.900692. Epub 2014 Apr 14. PMID 24730354
- [Background] Ho SS, Radavelli-Bagatini S, Dhaliwal SS, Hills AP, Pal S. Resistance, aerobic, and combination training on vascular function in overweight and obese adults. J Clin Hypertens (Greenwich). 2012 Dec;14(12):848-54. doi: 10.1111/j.1751-7176.2012.00700.x. Epub 2012 Aug 20. PMID 23205751
- [Background] Su L, Fu J, Sun S, Zhao G, Cheng W, Dou C, Quan M. Effects of HIIT and MICT on cardiovascular risk factors in adults with overweight and/or obesity: A meta-analysis. PLoS One. 2019 Jan 28;14(1):e0210644. doi: 10.1371/journal.pone.0210644. eCollection 2019. PMID 30689632